CLINICAL TRIAL: NCT03629496
Title: Developing an Arts-based Intervention for Patients With End-stage Kidney Disease Whilst Receiving Haemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Helen Noble, Chief Investigator, Lecturer, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B18-18
Record Dates: First submitted 2018-07-23; First posted 2018-08-14 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Feasibility Study; End Stage Renal Disease on Dialysis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Feasibility randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arts-based intervention (Experimental): Participants will participate in 6x1 hourly art sessions over a period of 3 weeks while they receive their haemodialysis treatment. This will involve 1:1 facilitation with a student and will involve visual arts including sketching, water colour painting and pen and ink, and creative writing activities. Participants will be provided with their own art supplies for infection control purposes and these will be kept on the unit in between sessions. Participants will have an option of displaying completed work in the reception area of the unit during their sessions.
  Interventions: Other: Arts-based intervention
- Control (No Intervention): Participants will receive usual care during their haemodialysis sessions and will be asked not to engage in any creative writing or visual arts during their haemodialysis sessions for the duration of the study. Once data collection has been completed the participants in the control group will receive art supplies and a single facilitated session on haemodialysis for the purpose of equity.

INTERVENTIONS:
Other: Arts-based intervention — 6x1 hourly facilitated art sessions during haemodialysis. Participants will be provided with an option of visual art or creative writing, the artistic materials used will include graphite pencils, colouring pencils, water colour paints and graphic pens. Participants will be provided with their own art supplies for infection control purposes. During each session participants will be allowed to self-select a subject matter or be provided with binary prompts to facilitate decision making. Participants will also have an option of displaying completed work in the reception area of the unit during their haemodialysis sessions.
  Arms: Arts-based intervention

SUMMARY:
This research study aims to develop an arts-based intervention for patients with end-stage kidney disease (ESKD) that can be implemented during haemodialysis sessions, and to assess the feasibility of a randomised controlled trial (RCT). Haemodialysis is the most common treatment for patients with ESKD; it involves attending hospital three times a week for a period of four hours each time, during that time the patient is connected to a dialysing unit that drains and filters their blood, performing the role of the damaged kidneys. Patients with ESKD receiving haemodialysis report low quality of life (QoL) and poor mental health. Arts-based interventions have been used in a variety of different settings to improve both QoL and mental health, but there's a lack of research assessing their effectiveness in patients with ESKD receiving haemodialysis.

This study will develop an arts-based intervention by reviewing the existing literature and forming an advisory group consisting of patients, healthcare staff, artists and academics. Once developed a feasibility RCT will be conducted on a haemodialysis unit. The feasibility RCT will involve establishing the recruitment, participation and retention rates of patients who are eligible for inclusion. A process evaluation will be conducted alongside the feasibility trial; this will involve interviews with patients and focus groups with staff to explore experiences of the intervention. Finally a feasibility economic evaluation will be conducted to explore methods for a cost-effectiveness analysis within an RCT. The hope is this study will contribute to a future RCT that will evaluate the impact of arts-based interventions on the QoL and mental health of patients receiving haemodialysis.

DETAILED DESCRIPTION:
This study consists of four phases and will utilise a mixed methods design. The first phase is the development of the intervention, the second phase is a feasibility randomised controlled trial (RCT), the third phase is a qualitative process evaluation and the fourth phase is a feasibility economic evaluation.

The first phase will involve the development of the intervention and will follow the development framework published by Fancourt in 'Arts in Health' (2017). This framework was developed specifically to inform arts-based interventions for healthcare contexts, and focuses primarily on identifying the needs of patients and staff within the clinical setting. The development will be informed by a systematic literature review and an interdisciplinary advisory group. The advisory group will consist of three patient representatives, two staff representatives from the haemodialysis unit, a renal counsellor from the Northern Health and Social Care Trust, two artist representatives from Arts Care Northern Ireland, the Chief Executive Officer from Arts Care Northern Ireland, the Community Wellbeing Manager in the Northern Health and Social Care Trust, a representative from the Renal Arts Group at Queen's, a representative from the University of Florida Arts in Medicine faculty, and a statistician. They will meet approximately every three months to inform the intervention and the research process.

The second phase will be a feasibility RCT that will involve recruiting 30 participants from Antrim Area Hospital's haemodialysis unit. Feasibility RCT's are necessary to determine whether a definitive randomised controlled trial can and should be conducted, and to identify the key areas within the methodology that work well or need to be adapted.

Recruitment will take place over seven months.Half the participants will be randomly allocated to the experimental group who will receive the intervention and half will be randomly allocated to the control group who will receive usual care.Participants will not be randomly allocated on an individual level, but instead will be randomly allocated according to the days of the week that they attend for haemodialysis. Patients receiving haemodialysis attend hospital on a set shift pattern, either Monday, Wednesday and Friday, or Tuesday, Thursday and Saturday. As the unit is open planned there is a risk that participants allocated to the control group will observe the intervention taking place if random allocation is done on an individual basis and this may influence the outcome; therefore randomisation will occur according to shift pattern to reduce the risk of contamination. The intervention will consist of an artistic activity that is minimally disruptive to the clinical setting, such as painting, sketching, pen and ink or creative writing. The intervention will be done at the bedside and will be adapted to ensure that vascular access is maintained. In order to ensure infection control protocols are followed each participant will receive their own set of art supplies to prevent the potential spread of infection through contaminated shared materials. The intervention will involve 6 sessions that will be administered over the course of 3 weeks for approximately an hour during dialysis sessions.

The third phase is the qualitative process evaluation. Participants will consist of both patients on the unit and staff who are working within the unit. Patients recruited will include those who have participated in phase two of the study, both in the intervention and control group. Semi-structured interviews will be conducted with 13 patients in order to capture a broad range of experiences with the intervention and the research process, including potential methods to make the intervention more accessible or engaging, experiences of being randomisation and participating in a control group, and reasons for retention of participants. 3 focus groups will be conducted with healthcare staff who have experienced the intervention on the unit. Due to the potential impact that arts-based interventions could have on the responsibilities of staff and the environment that they work in it is important to consider their experiences within the process evaluation as well, including identifying any barriers or facilitators to implementing the intervention in the dialysis setting.

Phase four is the feasibility economic evaluation. Participants who have been recruited into phase two of the study will be asked to complete a Patient Service Use Log throughout the study, this will be completed with the PhD student during the haemodialysis session, and the approximate cost of the intervention will be also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* Receiving haemodialysis
* Physically and cognitively able to consent and take part in art activities

Exclusion Criteria:

* Under 18
* Unable to read, write or speak English.
* Physically and cognitively unable to consent and take part in art activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention rates | Seven months
  Amount of participants recruited into the study, and the amount of the participants who remain in the study until its conclusion.

SECONDARY OUTCOMES:
Completion rate of Kidney Disease Quality of Life Short Form 36 | Data collection at baseline, 3 weeks, 6 weeks and 3 months per participant
  The Kidney Disease Quality of Life Short Form 36 (KDQoL-SF36) is a disease specific quality of life measure, where higher scores represent better self-reported quality of life. This will be administered to determine whether it is an appropriate outcome measure for a definitive trial as determined by completion rates, the proportion of recruited participants who complete the questionnaire. As this is a feasibility study and is not statistically powered to establish an effect the scores from the KDQOL-SF 36 will not be used for hypothesis testing.
Proportion of missing data from Kidney Disease Quality of Life Short Form 36 | Data collection at baseline, 3 weeks, 6 weeks and 3 months per participant
  The Kidney Disease Quality of Life Short Form 36 (KDQoL-SF36) is a disease specific quality of life measure, where higher scores represent better self-reported quality of life. This will be administered to determine whether it is an appropriate outcome measure for a definitive trial as determined by proportion of missing data from the 36 total items included in the scale, per participant. As this is a feasibility study and is not statistically powered to establish an effect the scores from the KDQOL-SF 36 will not be used for hypothesis testing.
Complete rate of missing data from Hospital Anxiety and Depression Scale | Data collection at baseline, 3 weeks, 6 weeks and 3 months per participant.
  The Hospital Anxiety and Depression scale (HADS) is a scale that detects depression, anxiety and emotional distress in hospitalised patients, where higher values indicate a worse outcome. It will be administered to determine whether it is an appropriate outcome measure for a definitive trial as determined by completion rates, the proportion of recruited participants who complete the questionnaire. As this is a feasibility study and is not statistically powered to establish an effect the scores from the HADS will not be used for hypothesis testing.
Proportion of missing data from Hospital Anxiety and Depression Scale | Data collection at baseline, 3 weeks, 6 weeks and 3 months per participant.
  The Hospital Anxiety and Depression scale (HADS) is a scale that detects depression, anxiety and emotional distress in hospitalised patients, where higher values indicate a worse outcome. It will be administered to determine whether it is an appropriate outcome measure for a definitive trial as determined by proportion of missing data from the 14 total items included in the scale, per participant. As this is a feasibility study and is not statistically powered to establish an effect the scores from the HADS will not be used for hypothesis testing.
Completion rate of EuroQuol 5d 5l (EQ-5d-5l) | Data collection at baseline, 3 weeks, 6 weeks and 3 months per participant
  EuroQuol-5D-5L (EQ-5D-5L) is a standardised measure of health-related quality of life commonly used in economic evaluations to calculate cost-utility. The EQ-5D-5L will be administered to determine whether it is an appropriate outcome measure for a definitive trial (specifically for an economic evaluation) as determined by completion rates, the proportion of recruited participants who complete the questionnaire. As this is a feasibility study and is not statistically powered to establish an effect the scores from the EQ-5D-5L will not be used to calculate cost-utility of the intervention.
Proportion of missing data from EuroQuol 5d 5l (EQ-5d-5l) | Data collection at baseline, 3 weeks, 6 weeks and 3 months per participant
  EuroQuol-5D-5L (EQ-5D-5L) is a standardised measure of health-related quality of life commonly used in economic evaluations to calculate cost-utility. The EQ-5D-5L will be administered to determine whether it is an appropriate outcome measure for a definitive trial (specifically for an economic evaluation) as determined by proportion of missing data from the 6 total items included in the scale. As this is a feasibility study and is not statistically powered to establish an effect the scores from the EQ-5D-5L will not be used to calculate cost-utility of the intervention.
Completion rate of Patient Service Use Log | Data collection at baseline, 3 weeks, 6 weeks and 3 months per participant
  A Patient Service Use Log will be administered to determine whether it is an appropriate method to capture healthcare resource use data for an economic evaluation within a definitive trial as determined by completion rates , the proportion of recruited participants who complete the log. As this is a feasibility study and is not statistically powered to establish an effect the data from the Patient Resource Use log will not be used to calculate cost-utility of the intervention.
Proportion of missing data from Patient Service Use Log | Data collection at baseline, 3 weeks, 6 weeks and 3 months per participant
  A Patient Service Use Log will be administered to determine whether it is an appropriate method to capture healthcare resource use data for an economic evaluation within a definitive trial as determined by proportion of missing data per participant. As this is a feasibility study and is not statistically powered to establish an effect the data from the Patient Resource Use log will not be used to calculate cost-utility of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Noble, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Antrim Area Hospital Renal Unit, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carswell C, Reid J, Walsh I, Johnston W, McAneney H, Mullan R, Lee JB, Nelson H, Matthews M, Weatherup E, Spencer A, Michelo J, Quail A, Kielty G, Mackenzie A, Elliott J, Arbuckle N, Wilson A, Noble H. A mixed-methods feasibility study of an arts-based intervention for patients receiving maintenance haemodialysis. BMC Nephrol. 2020 Nov 19;21(1):497. doi: 10.1186/s12882-020-02162-4. PMID 33213413
- [Derived] Carswell C, Reid J, Walsh I, McAneney H, Noble H. Implementing an arts-based intervention for patients with end-stage kidney disease whilst receiving haemodialysis: a feasibility study protocol. Pilot Feasibility Stud. 2019 Jan 5;5:1. doi: 10.1186/s40814-018-0389-y. eCollection 2019. PMID 30622728

DOCUMENTS (3):
  • Study Protocol (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03629496/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT03629496/SAP_001.pdf
  • Informed Consent Form (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT03629496/ICF_002.pdf